CLINICAL TRIAL: NCT02688335
Title: Home-Use Impact and Effectiveness of Cloud 9
Acronym: Cloud9
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00052615
Record Dates: First submitted 2016-02-12; First posted 2016-02-23 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Snoring
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cloud9 Snoring Treatment (Experimental): Snoring participants will be instructed to use the device as much as possible for 2 weeks.
  Interventions: Device: Cloud9

INTERVENTIONS:
Device: Cloud9 — Low-pressure Continuous Positive Airway Pressure (CPAP = 2 - 4 cm H2O).
  Other Names: inSleep Technologies

SUMMARY:
This is an interventional study in which patients with a history of habitual snoring will use the low-pressure CPAP device at home for about 4 weeks. This study is designed to document the adherence of the snorer, the acceptance and comfort of the therapy, and bed partners' subjective report of improvement in sleep quality, and/or reduction or elimination of snoring. Study outcomes will consist of an assessment of the nightly usage time, and questionnaires that the snorer and the bed-partner have to complete before the start of the study and at the end of the study period.

DETAILED DESCRIPTION:
This is an interventional study in which patients with a history of habitual snoring use the Cloud9™ Continuous Positive Airway Pressure (CPAP) device that delivers a low level of continuous nasal air pressure between 2 cm H2O and 4 cm H2O, for about four weeks at their home. This study is designed to document the adherence of the snorer, the acceptance and comfort of the therapy, and bed partners' subjective report of improvement in sleep quality, and/or reduction or elimination of snoring.

Study Procedures

Study Procedures

Baseline Assessment: The study begins with a baseline assessment to determine whether each participant meets the entry criteria for the study. After consent, participant snorers will have a history and physical exam to confirm entry criteria and answer questionnaires: Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Snore Outcomes Survey (SOS), and Stanford Sleepiness Scale (SSS) to assess their sleepiness and snoring. In a second step, snoring participants who initially meet the entry criteria will receive a full night Home Sleep Test (HST) to confirm snoring and to rule out sleep apnea or any other sleep related disorder. Participants who already performed a full night polysomnography (PSG) as a part of the earlier sleep lab study for the Cloud9 device (Treatment of Snoring NA_00073250) do not have to be re-screened, if the earlier PSG is not older than 36 months, and the participant's BMI remains within 3 kg/m2 of its original value. In parallel, the snorer's bed-partner will be asked to complete baseline questionnaires: ESS, PSQI, Spouse/Bed-partner Survey (SBPS), and supplement, SSS, and snore assessment according to Visual Analog Scale (VAS).

Baseline Week: Snorers and bed-partners will be asked to wear Actigraphy watches for approximately one-week prior to the initiation of treatment at home with the study device.

Home-Trial: At the end of the baseline week, snoring participants will be asked to use the device at home for 4 weeks. Usage data will be recorded by a power logger and read when returned to the study site at the end of study. Snoring participants will receive a study coordinator call on the day after night 1 of the home trial. Additionally, snoring participants will receive a coordinator call weekly thereafter, to assess the user experience with the device. Snorers and bed-partners will continue to wear Actigraphy monitors throughout the home-trial.

Final Visit: At the end of the 4 weeks of home use, participants will return all study equipment to the sleep lab. Usage data from the data logger will be read for compliance rates. Snoring participants and their bed partners will also complete a final set of questionnaires as before (ESS, PSQI, SOS, SBPS and supplement. Bed partners will rate snoring using VAS. Snorers will also be asked to complete a Comfort and Acceptability Survey and the Sleep Apnea Quality of Life Index (SAQLI) Treatment related questions.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 18 years of age.
* Patient is willing and able to provide written Informed Consent utilizing a Patient Information and Consent form that has been reviewed and approved by a governing Institutional Review Board (IRB).
* Patient has a bed partner willing to participate in the study
* Patient has a history of habitual snoring (almost every night or every night) as determined by a bed-partner; bed-partner subjectively reports that snoring is a considerable burden for her/him.
* Patient has been pre-screened and demonstrates an Epworth Questionnaire (an assessment of daytime sleepiness; high number = greater sleepiness) score of less than 11, no history of witnessed apneas or nocturnal gasping/choking episodes and a BMI ≤ 35, or subjects with a BMI >35 who have no significant sleep apnea already documented on an overnight sleep study.

Exclusion Criteria: (For subjects recruited from the previous inSleep protocol, the BMI must be in a range of ±3 kg/m2 of the earlier recorded value)

* Patient has been diagnosed with Chronic Obstructive Pulmonary Disease (COPD), asthma, emphysema or chronic bronchitis.
* Patient has a history of heart disease, heart attack or stroke.
* Patient has uncontrolled or poorly controlled hypertension.
* Patient has been diagnosed with Obstructive Sleep Apnea (OSA), defined as Apnea-Hypopnea Index (AHI) ≥ 15. Hypopnea is defined as a discernible reduction in flow that is associated with a greater than or equal to 4% desaturation.
* Pregnancy of the snoring participant, by self-report. If there is any doubt concerning status, a urine pregnancy test will be performed.
* Patient is currently participating in another clinical study for which follow-up is ongoing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Snoring Severity | 1 night
  Snoring intensity will be assessed from standard polysomnography (if completed during previous trial), otherwise a WatchPAT device will be used at home for one night to measure sleep and snoring. The WatchPAT is a watch-like device worn on the wrist, which includes finger sensor to monitor oxygen saturation.
Bed Partner Sleep Quality - Actigraphy | 4 weeks
  This will be assessed via activity monitoring measured by Actigraphs worn on the wrist.

SECONDARY OUTCOMES:
Usage Time of the Cloud9 device | 4 weeks
  The Cloud9 device will be connected to a power logger and data collected at the end of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Alan R Schwartz, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview - Asthma and Allegy Building, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with researchers outside the primary research group for secondary purposes.